CLINICAL TRIAL: NCT06343727
Title: A High Protein Egg White Pudding for People With Kidney Failure (HiPE KF)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seven Oaks Hospital Chronic Disease Innovation Centre (Network)
Collaborators: University of Manitoba (Other); Manitoba Egg Farmers (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS25870 (H2023:026)
Record Dates: First submitted 2024-02-07; First posted 2024-04-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Kidney Failure; Frailty; Kidney Disease, Chronic
MeSH Terms: conditions — Renal Insufficiency; Frailty; Renal Insufficiency, Chronic | interventions — Ensure Plus

STUDY DESIGN:
Intervention Model Description: This trial is an open-label randomized controlled parallel arm feasibility trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Egg white protein pudding (Experimental): Participants will receive egg white pudding at the end of their dialysis treatments 3-days per week.
  Interventions: Dietary Supplement: Egg white protein pudding
- : Standard dietary supplement (Active Comparator): Participants will receive Ensure Plus at the end of their dialysis treatments 3-days per week.
  Interventions: Dietary Supplement: : Ensure Plus

INTERVENTIONS:
Dietary Supplement: Egg white protein pudding — Will consume one egg white protein pudding at the end of their dialysis treatments 3-days per week for 12 weeks
  Arms: Egg white protein pudding
Dietary Supplement: : Ensure Plus — Will consume one Ensure Plus at the end of their dialysis treatments 3-days per week for 12 weeks
  Arms: : Standard dietary supplement

SUMMARY:
The goal of this clinical trial is to compare protein supplements in patients with kidney failure on dialysis. The main questions it aims to answer are:

* To determine whether the supplementation of egg white protein pudding in a population of individuals with kidney failure on dialysis is feasible.
* To determine whether egg white protein pudding supplementation improves serum albumin similar to other standard nutritional supplements.
* To determine the effects of the egg white protein pudding on frailty measures, dietary intakes and analytes in the blood. Participants will receive either the egg white pudding (experimental) or control (Ensure plus) at the end of their dialysis treatments 3-days per week for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial
* Male or female aged ≥18 years with CKD
* On chronic in-center hemodialysis for > 3 months
* Serum albumin <35 g/L
* No expected change in dialysis modality or relocation outside of Winnipeg during the intervention period (12 weeks)

Exclusion Criteria:

* Allergy to eggs
* History of renal transplant
* Serum albumin ≥ 35 g/L
* Bowel diseases
* Cancer
* Pregnancy
* Receiving chemotherapy treatment
* Inability to consume treatment product
* Allergy to study treatment ingredients
* Planning on starting an exercise program during the duration of the trial
* Inability to obtain written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Eligibility to randomization ratio | Measured at the end of 12 weeks.
  A ratio of eligibility to randomization will be collected at 12 months using pre-specified red-yellow-green progression criteria to investigate egg pudding intervention feasibility. The trial will be considered feasible if ratio falls within green zone (>0.5). The outcome in the yellow zone (0.2-0.5) indicate that modifications to trial design may be necessary and in the red zone (<0.2) will suggest the trial is not feasible.
Recruitment rate | 12 months
  Recruitment rate will be assessed as the number of new participants enrolled per site per month during active recruitment using the red-yellow-green progression criteria.
  Green: ≥ 0.75 participants/site/month - Feasible; Yellow: 0.25 - <0.75 participants/site/month - Modification may be necessary; Red: < 0.25 participants /site/month - Not feasible
Follow up rate | Measured at the end of 12 weeks.
  Follow-up rate (% of participant outcomes) will be calculated using the red-yellow-green progression criteria.
  Green: > 90% - Feasible; Yellow: (75% - 90%) -Modifications may be necessary; Red: <75% -Not feasible.
Adherence to Intervention | Measured at the end of12 weeks
  Adherence to egg white product intervention (% of dispensed egg white protein consumed) will be calculated using red-yellow-green progression criteria.
  Green: > 75% - Feasible; Yellow: 50%-75% - Modifications may be necessary; Red: <50% - Not feasible

SECONDARY OUTCOMES:
Hand grip strength | Measured at the end of 12 weeks.
  Measuring the amount of static force that the hand can squeeze around a dynamometer. Measured in kilograms and pounds.
Change in gait speed | Measured at the end of 12 weeks.
  Gait speed is measured by the predetermined distance/time to walk that distance (e.g., 5m/__sec)
Five rep chair stand time | Measured at the end of 12 weeks.
  the amount of time it takes for a participant to get up out of a chair five times measured in seconds
Tandem balance time | Measured at the end of 12 weeks.
  Measured in Seconds
Serum albumin | Measured at the end of 12 weeks.
  Serum albumin is measured in grams per deciliter (g/dL)
Serum bicarbonate | Measured at the end of 12 weeks.
  Serum bicarbonate concentration in milliequivalents per liter (mEq/L)
Calcium | Measured at the end of 12 weeks.
  Total blood calcium concentration in mmol/L
chloride | Measured at the end of 12 weeks.
  Total blood chloride concentration in mmol/L
phosphorus | Measured at the end of 12 weeks.
  The total blood phosphorus concentration in mmol/L
Potassium | Measured at the end of 12 weeks.
  The total blood potassium concentration in mmol/L
Sodium | Measured at the end of 12 weeks.
  The total sodium concentration in mmol/L
HbA1c | Measured at the end of 12 weeks.
  Total blood glucose concentration in mmol/L
Dry Weight | Measured at the end of 12 weeks
  Measured in kg
Height | Measured at the end of 12 weeks
  Measured in cm
Pre-dialysis Blood pressure | Measured at the end of 12 weeks
  Systolic and diastolic blood pressure measured in mmHg

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Seven Oaks General Hospital, Winnipeg, Manitoba
  - Health Science Centre, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No